CLINICAL TRIAL: NCT04491188
Title: Plasma Amino Acid Response to Whey Protein Ingestion Following 28-days of Probiotic (Bacillus Subtilis DE111) Supplementation in Active Men and Women
Brief Title: Plasma Amino Acid Response to Whey Protein Ingestion Following 28-days of Probiotic Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lipscomb University (Other)
Collaborators: Deerland Enzymes (Industry)
Responsible Party: Principal Investigator, Jeremy Townsend, Assistant Professor, Lipscomb University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 01082018
Record Dates: First submitted 2020-07-20; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Focus of Study is Amino Acid Appearace in Blood

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): 1 x10-9 CFU Bacillus subtilis DE111 was consumed daily for 28-days
  Interventions: Dietary Supplement: Bacillus subtilis DE111
- Placebo (Placebo Comparator): Maltodextrin placebo was consumed for 28-days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bacillus subtilis DE111 — 1 x10-9 CFU Bacillus subtilis DE111 probiotic
  Arms: Probiotic
Dietary Supplement: Placebo — Maltodextrin placebo
  Arms: Placebo

SUMMARY:
Active males and females consumed a probiotic for 28-days. Before and after the intervention period, participants reported to the lab in a fasted state where they consumed 25 grams of whey protein. Following drink consumption, participants provided blood draws at 15-minute intervals. Blood samples were analyzed for amino acid concentrations.

ELIGIBILITY:
Inclusion Criteria:

* 18-34 years old Participants must have at least 1 year of resistance training experience.
* Free of any physical limitations, medications, and supplements that may affect performance, as determined by a health and activity questionnaire.
* Are free of musculoskeletal injuries
* Are not taking medications that may interfere with study measurements

Exclusion Criteria:

* Taking any other nutritional supplement or performance enhancing drug.
* Any chronic illness that causes continuous medical care
* Taking any other nutritional supplement or performance enhancing drug.
* Any chronic illness that causes continuous medical care.

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-03 (Actual)

PRIMARY OUTCOMES:
Plasma Amino Acid response | 28-days
  We measured plasma amino acid concentrations before and after the 28-day intervention

SECONDARY OUTCOMES:
Body Composition | 28-days
  Body Fat Percentage (%) will be monitored before and after the intervention via Bioelectical Impedance Analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Jeremy Townsend, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided